CLINICAL TRIAL: NCT03967938
Title: Efficacy of Olaparib in Advanced Cancers Occurring in Patients With Germline Mutations or Somatic Tumor Mutations in Homologous Recombination Genes
Acronym: 1-2018 BSMO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AZ-VUB (Other)
Collaborators: AstraZeneca (Industry); Kom Op Tegen Kanker (Other)
Responsible Party: Principal Investigator, Dr. Sofie Joris, Coordinator Investigator, AZ-VUB
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Precision 2 - Olaparib
Record Dates: First submitted 2019-02-11; First posted 2019-05-30 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Advanced Cancers Harbouring Mutations in HRG
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Olaparib (Experimental): tablets of 300mg twice daily until disease progression
  Interventions: Drug: Olaparib Oral Capsule

INTERVENTIONS:
Drug: Olaparib Oral Capsule — Olaparib tablets 300mg twice daily

SUMMARY:
At present targeted therapy with the PARP inhibitor olaparib has become standard of care in advanced platinum sensitive BRCA1/2 mutant ovarian cancer. The key in this sensitivity is the loss of homologous recombination (HR) function. The current project aims to treat patients with any type of cancer carrying in their germline a mutation in genes that generate such an homologous recombination deficiency (HRD) or have an acquired somatic mutation in their tumor with the targeted PARP inhibitor olaparib. The project would thus bring access to a targeted drug matched to the genomic profile of the tumor of these patients and provide oncologists with information regarding efficacy and safety of olaparib in these patients. This evidence could then later lead to a more routine regulatory access.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Female or male aged > 18 years
3. Histologically proven advanced cancer, either locally or metastatic, harboring a specific pathogenic genetic alteration (with the exception of breast, pancreas, or prostate cancer patients harboring a BRCA1/2 mutation and HRD ovarian cancer)
4. No approved targeted therapy for the specific genetic alteration in the specific tumor type
5. No other genomic driven phase I, II or III trial available for the specific genomic alteration in the specific tumor type
6. Available tumor tissue for verification of the mutation by Sanger sequencing.
7. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment.
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
9. Patients must have a life expectancy ≥16 weeks
10. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.
11. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
12. At least one lesion (measurable and/or non-measurable) that can be accurately assessed at baseline by CT and is suitable for repeated assessment.
13. *Formalin fixed, paraffin embedded (FFPE) tumour sample from the primary cancer must be available for local genetic testing.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Ovarian cancer patients harboring a HRD and breast, prostate and pancreas cancer patients who carry a BRCA1/2 mutation
3. Previous enrolment in the present study
4. Participation in another clinical study with an investigational product during the last 4 weeks or radiotherapy (except for palliative reasons) within three weeks prior to study treatment.
5. History of non-compliance to medical regimens
6. Any previous treatment with PARP inhibitor, including olaparib.
7. Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma, or other solid tumours including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥5 years. Patients with a history of localized triple negative breast cancer may be eligible, provided they completed their adjuvant chemotherapy more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
8. Resting ECG with QTc > 470 msec on 2 or more time points within a 24 hour period or indicating uncontrolled, potentially reversible cardiac conditions as judged by the investigator (er., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500ms, electrolyte disturbances, etc.) or patients with congenital long QT syndrome
9. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within four weeks prior to study treatment. Patients must have recovered from radiotherapy toxicities prior to enrollment.
10. Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
11. Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
12. Persistent toxicities (Common Terminology Criteria for Adverse Event (CTCAE) > grade 2) caused by previous cancer therapy, excluding alopecia.
13. Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
14. Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
15. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
16. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
17. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
18. Breast feeding women. (delete if male population)
19. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
20. Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
21. Patients with known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids
22. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
23. Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable, for timing refer to inclusion criteria no.3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2019-02-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Response rate according to RECIST 1.1 | every 2 months from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  The primary analysis will estimate the proportion of patients who achieve confirmed objective response according to the RECIST criteria. Objective response is defined as confirmed CR or PR.
Response duration according to RECIST 1.1 | from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Patients whose best RECIST assessment is stable disease, partial, or complete response will be considered to have achieved disease control. Descriptive statistics will be produced for the duration of confirmed objective response and disease control.

SECONDARY OUTCOMES:
locus-specific LOH | through study completion, an average of 1 year
  Correlate efficacy with locus-specific LOH in the tumors in case of cancers atypical for the germline mutations
PFS | every 2 months from date of randomization until teh date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  PFS is the time from start of treatment until the occurrence of disease progression or death, whichever comes first. Date of progression is the earliest of (1) date of imaging showing disease progression, or (2) date of investigator assessment of clinical progression, or (3) date recorded from post study follow-up for disease progression, or (4) start of new anti-cancer treatment (i.e., either the secondary treatment regimen or other anti-cancer treatment).
OS | every 2 months from date of randomization until teh date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  OS is the time from start of treatment until death, for whatever reason.

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Joris, Dr, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No